CLINICAL TRIAL: NCT02314962
Title: Diagnostic and Clinical Accuracy of Integrated Magnetic Resonance Imaging and Computed Tomography Perfusion in PET/MRI in Comparison to PET/CT in Solid Tumors
Brief Title: PET/MRI Perfusion and CT Perfusion in Solid Tumors
Acronym: Perfusion
Status: Terminated | Type: Observational
Why Stopped: Slow enrolment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK ZH Nr 20140077
Record Dates: First submitted 2014-10-23; First posted 2014-12-11 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: CT Perfusion and MRI Perfusion in Solid Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diagnostic comparison between PET/CT and PET/MRI with integrated perfusion measurement in CT and MR. Study aim is to gain knowledge about additional value of CT perfusion and MR perfusion in solid tumors concerning tumor physiology, diagnostic accuracy and possibly prognostic.

ELIGIBILITY:
Inclusion Criteria:

* indication as stated above
* written informed consent
* patients with suspected or confirmed solid malignant tumors of the neck, chest or abdomen who have an indication for a PET/CT

Exclusion Criteria:

* pregnant or breast feeding women
* non compliance of the patient to follow the study instructions (e.g. hearing problems, dementia)
* Inclusion in another clinical trial 30 days prior to inclusion
* age < 30years
* contraindication for MRI (cardiac pacemaker, certain metal implants, claustrophobia
* known allergies to contrast CT or MRI contrast media
* patients with an glomerular filtration rate of < 60ml/min/1.73m2

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed solid malignant tumors of the neck, chest or abdomen who have an indication for a PET/CT
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement of blood flow, blood volume and transfer constant (Ktrans) with CT-Perfusion and PET/MR-perfusion in solid tumors. | 18 months

SECONDARY OUTCOMES:
Correlation of blood flow, blood volume and transfer constant (Ktrans) measured with CT-Perfusion and PET/MR-perfusion with progression free survival in solid tumors. | 18 months

OTHER OUTCOMES:
Measurement of blood flow (mL/100 mg tissue/min) with CT-Perfusion and PET/MR-perfusion in solid tumors. | 18 months
Measurement of blood volume (mL/100 mg tissue) with CT-Perfusion and PET/MR-perfusion in solid tumors. | 18 months
Measurement of transfer constant with PET/MR-perfusion in solid tumors. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Hospital Zurich, Diagnostic and Interventional Radiology
Locations (1):
- University Hospital Zurich, Diagnostic and Interventional Radiology, Zurich, Canton of Zurich, Switzerland